CLINICAL TRIAL: NCT06637397
Title: Assessing the Safety and Effectiveness of Weizmania Coagulant BC99 in Relieving Functional Constipation in Adults Based on Randomized, Double-Blind, Placebo-Controlled Trials
Brief Title: Probiotics for Alleviating Functional Constipation in Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WK2024007
Record Dates: First submitted 2024-05-27; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-04

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic Group (Experimental): Participants receive one sachet per day containing probiotic BC99 and maltodextrin (Week 0 to Week8).
  Interventions: Dietary Supplement: Probiotic
- Placebo Group (Placebo Comparator): Participants receive one sachet per day containing maltodextrin only, serving as the placebo(Week 0 to Week8).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — During the intervention, participants can consume BC99 daily and any adverse reactions were noted. Stool and serum samples were collected for analysis of 16S rRNA and serum inflammatory markers. Changes in intestinal flora and inflammatory factors before and after supplementation were assessed.
  Arms: Probiotic Group
Dietary Supplement: Placebo — During the intervention, participants can consume maltodextrin daily and any adverse reactions were noted. Stool and serum samples were collected for analysis of 16S rRNA and serum inflammatory markers. Changes in intestinal flora and inflammatory factors before and after supplementation were assessed.
  Arms: Placebo Group

SUMMARY:
To investigate the clinical effects of probiotics in relieving chronic constipation in adults, and evaluate the improvement of symptoms in patients with constipation as well as their impacts on gastrointestinal function, immunity, and gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese adults who meet the diagnostic criteria of Rome III, aged between 18 and 70;
2. Patients with chronic constipation (disease duration exceeding 6 months, with fewer than 3 bowel movements per week and/or Bristol stool form scale types 1 and 2);
3. Able to complete the study according to the requirements of the experimental protocol;
4. Patients who have signed the informed consent form;
5. Research participants (including male participants) who do not have fertility plans from 14 days before screening to 6 months after the end of the trial and are willing to take effective contraceptive measures voluntarily.

Exclusion Criteria:

1. Individuals who have taken items with similar functions to the tested product within a short period of time, which may affect the judgment of the results;
2. Patients who have changed their diet during the study period;
3. Patients with severe allergies and immune deficiencies;
4. Female patients who are pregnant, breastfeeding, or have plans to become pregnant;
5. Patients with severe diseases in vital organs such as cardiovascular, lung, liver, and kidney, as well as severe metabolic diseases such as diabetes, thyroid disease, malignant tumors, and severe immune system diseases;
6. Individuals who have used antibiotics within the past two weeks;
7. Individuals with severe psychological or mental illnesses;
8. Participants who have not consumed the tested samples as required or failed to follow up on time, resulting in an inability to determine the effectiveness;
9. Other research participants deemed unsuitable for participation by the researchers.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Assessing the Improvement of Chronic Constipation Symptoms Following Probiotic Intervention. | 8 weeks
  Constipation symptoms are measured using Bristol Stool Form Scale (BSFS).

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Henan University of Science and Technology, Luoyang, Henan
  - The School of Food and Bioengineering, Henan University of Science and Technolog, Luoyang, Henan

IPD SHARING:
Plan to Share IPD: No